CLINICAL TRIAL: NCT01050205
Title: Diabetes Prevention Translation Project: the Healthy Lifestyle Project
Brief Title: Diabetes Prevention Translation: the Healthy Lifestyle Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Andrea Kriska, PhD, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO10010131; R18DK081323-04 (NIH)
Record Dates: First submitted 2010-01-13; First posted 2010-01-15 (Estimated); Results first posted 2017-07-25 (Actual); Last update posted 2017-08-25 (Actual); Status verified 2017-07

CONDITIONS: Diabetes; Cardiovascular Risk Factor
Keywords: Diabetes Prevention; Cardiovascular Risk Reduction; Lifestyle Intervention; Group Lifestyle Balance
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Current Intervention (Active Comparator): Eligible participants will be asked to choose Group Lifestyle Balance Group (GLB-Group) or Group Lifestyle Balance DVD (GLB-DVD). Upon choosing, participants will be randomly assigned to "Current intervention" Arm in which case they will receive the intervention immediately.
  Interventions: Behavioral: Current Intervention
- Delayed Intervention (Active Comparator): Eligible participants will be asked to choose Group Lifestyle Balance Group (GLB-Group) or Group Lifestyle Balance DVD (GLB-DVD). Upon choosing, participants will be randomly assigned to "Delayed Intervention" Arm in which case they will receive delayed intervention at 6 months.
  Interventions: Behavioral: Delayed Intervention

INTERVENTIONS:
Behavioral: Current Intervention — Participants assigned to Current Intervention will receive the intervention described below immediately after randomization. The one-year GLB program is an adaptation of the successful DPP lifestyle intervention. The goals of the intervention are to achieve and maintain a 7% weight loss, and to safely and progressively increase physical activity to 150 minutes per week of moderately intense physical activity.
  GLB-GROUP: group meetings weekly transitioning to monthly over one year led by a trained coach. GLB-DVD: Consists of a series of taped sessions of a staged GLB group following a script which was developed to closely follow the GLB program. GLB-DVD participants complete the sessions via DVD and have telephonic contact with their coach as well as monthly group meetings.
  Arms: Current Intervention
Behavioral: Delayed Intervention — Participants assigned to Delayed Intervention receive the same intervention as Current Intervention Group, 6 months from randomization. The one-year GLB program is an adaptation of the successful DPP lifestyle intervention. The goals of the intervention are to achieve and maintain a 7% weight loss, and to safely and progressively increase physical activity to 150 minutes per week of moderately intense physical activity.
  GLB-GROUP: group meetings weekly transitioning to monthly over one year led by a trained coach. GLB-DVD: Consists of a series of taped sessions of a staged GLB group following a script which was developed to closely follow the GLB program. GLB-DVD participants complete the sessions via DVD and have telephonic contact with their coach as well as monthly group meetings.
  Arms: Delayed Intervention

SUMMARY:
The Diabetes Prevention Program (DPP), a large research study conducted in the United States, found that lifestyle intervention was effective in lowering risk for development of type 2 diabetes. It is important to evaluate the DPP lifestyle interventions in "real world" settings. The purpose of this project is to test an adapted version of the DPP lifestyle intervention in several community settings, including a worksite, a health care facility (primary care practice and local community centers dedicated to older adults.

DETAILED DESCRIPTION:
Evidence that lifestyle intervention can prevent or delay the development of type 2 diabetes has been demonstrated in several clinical trials including a multi center clinical trial in the US, the Diabetes Prevention Program (DPP). The challenge for public health is to translate this promising and proven behavioral intervention utilized in the DPP research effort to the "real world", i.e., how to make it work in diverse communities in a variety of local settings at a reduced cost so that the maximal number of those at risk can benefit.

The purpose of this application is to test a framework for translation of the DPP that includes: 1) demonstration of a training model for community health care professionals that includes initial training, support, and supervision in the delivery of a diabetes prevention curriculum and the needed behavioral lifestyle materials both initially and over time; 2) evaluation of a more compact and flexible DPP intervention program administered to each participant in a version of his or her choice (standard face-to-face group format or a DVD version of the same lifestyle intervention program content). These lifestyle intervention programs will be carried out in three different community settings; i.e. a health care practice, a worksite, and local centers in the community dedicated to healthy aging for older adults. Lastly, the cost-effectiveness analyses of the GLB intervention program in each of the three community settings will be tested.

ELIGIBILITY:
Inclusion Criteria:

* Screening Eligibility Criteria: Non-diabetic men and women from the specific study sites in the local area who are age 18 years and older at the time of screening with a BMI of at least 25 kg/m2 are eligible for screening.
* Intervention Eligibility Criteria: Individuals attending screening who are found to have prediabetes AND/OR metabolic syndrome are eligible to participate in the intervention. Pre-diabetes is defined as having a fasting glucose >100 mg/dL and <126mg/dL. Metabolic syndrome is defined as having at least 3 of the 5 following risk factors:

  1. Waist circumference (>40 inches men, >35 inches women);
  2. Blood pressure >130 mmHg (systolic) or >85 mmHg (diastolic) OR history of diagnosed hypertension
  3. Low HDL level (<40mg/dL men, <50 mg/dL women)
  4. Elevated triglyceride level >150 mg/dL
  5. Fasting glucose >100mg/dL and <126mg/dL All individuals enrolled in the study should have at least 6th grade reading/writing ability.

Exclusion Criteria:

* Screening Exclusionary Criteria: Women who are currently (or within past 6-weeks) pregnant or lactating, or any individual planning to leave the area before the end of the effort will be considered ineligible to participate in the screening.
* Intervention Exclusionary Criteria: Exclusionary criterion for intervention is the same as for screening. In addition, individuals who are on metformin or are identified as having diabetes as a result of the screening are not eligible. Individuals who have recently (within the past 3 months) initiated or changed their dosage of any blood pressure or lipid medication will also be excluded as being on an unstable regimen will complicate the interpretation of any blood pressure or lipid effects of the intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2010-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea M Kriska, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Kramer MK, Agee SC, Miller RG, Arena VC, Vanderwood KK, Eaglehouse YL, Venditti EM, Kriska AM. Translating the Diabetes Prevention Program Lifestyle Intervention to the Military Setting. Mil Med. 2023 May 16;188(5-6):1036-1045. doi: 10.1093/milmed/usac037. PMID 35234887
- [Derived] Devaraj SM, Napoleone JM, Miller RG, Rockette-Wagner B, Arena VC, Mitchell-Miland C, Saad MB, Kriska AM. The role of Sociodemographic factors on goal achievement in a community-based diabetes prevention program behavioral lifestyle intervention. BMC Public Health. 2021 Oct 2;21(1):1783. doi: 10.1186/s12889-021-11844-z. PMID 34600527
- [Derived] Rockette-Wagner B, Miller RG, Eaglehouse YL, Arena VC, Kramer MK, Kriska AM. Leisure Sedentary Behavior Levels and Meeting Program Goals in a Community Lifestyle Intervention for Diabetes Prevention. J Phys Act Health. 2021 Jan 1;18(1):44-51. doi: 10.1123/jpah.2020-0052. Epub 2020 Dec 22. PMID 33361473
- [Derived] Schafer GL, Songer TJ, Arena VC, Kramer MK, Miller RG, Kriska AM. Participant food and activity costs in a translational Diabetes Prevention Program. Transl Behav Med. 2021 Mar 16;11(2):351-358. doi: 10.1093/tbm/ibaa031. PMID 32298445
- [Derived] Kramer MK, Vanderwood KK, Arena VC, Miller RG, Meehan R, Eaglehouse YL, Schafer G, Venditti EM, Kriska AM. Evaluation of a Diabetes Prevention Program Lifestyle Intervention in Older Adults: A Randomized Controlled Study in Three Senior/Community Centers of Varying Socioeconomic Status. Diabetes Educ. 2018 Apr;44(2):118-129. doi: 10.1177/0145721718759982. Epub 2018 Mar 7. PMID 29514568
- [Derived] Eaglehouse YL, Rockette-Wagner B, Kramer MK, Arena VC, Miller RG, Vanderwood KK, Kriska AM. Physical Activity Levels in a Community Lifestyle Intervention: A Randomized Trial. Transl J Am Coll Sports Med. 2016 Jun 1;1(5):45-51. PMID 27551690
- [Derived] Eaglehouse YL, Schafer GL, Arena VC, Kramer MK, Miller RG, Kriska AM. Impact of a community-based lifestyle intervention program on health-related quality of life. Qual Life Res. 2016 Aug;25(8):1903-12. doi: 10.1007/s11136-016-1240-7. Epub 2016 Feb 20. PMID 26896960
- [Derived] Vanderwood KK, Kramer MK, Miller RG, Arena VC, Kriska AM. Evaluation of non-invasive screening measures to identify individuals with prediabetes. Diabetes Res Clin Pract. 2015 Jan;107(1):194-201. doi: 10.1016/j.diabres.2014.06.003. Epub 2014 Jun 21. PMID 25441924

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Individuals were recruited via screenings in 3 community settings: a) a local work site, b) 3 community/senior centers, and c) a military medical facility. The military medical facility was a pre-post study not an RCT. Results are presented for the RCT sites. Recruitment at these sites began in Fall of 2010 and was completed in Winter of 2013.
Groups:
- Current Intervention: At enrollment, participants randomly assigned to "Current Intervention" will receive the intervention immediately.The intervention is based on the Diabetes Prevention Program's successful lifestyle intervention with goals of achieving a 7% weight loss, and progressively increasing physical activity to 150 minutes per week of moderately intense physical activity.Participants will choose one of the following interventions:
  GLB-GROUP: Individuals who choose group delivery will attend weekly in-person group meetings for 12 weeks, then transition to bi-weekly and monthly meetings. GLB-DVD: Consists of a series of taped sessions of a staged GLB group following a script which was developed to closely follow the original Group Lifestyle Balance. Participants in GLB-DVD will also be invited to attend monthly group meetings and will receive weekly telephone calls from a trained coach.
- Delayed Intervention: At enrollment, participants randomly assigned to "Delayed intervention" will receive the intervention in 6 months. The intervention is identical to that received by participants assigned to the Current Intervention Arm and is based on the Diabetes Prevention Program's successful lifestyle intervention with goals of achieving a 7% weight loss, and progressively increasing physical activity to 150 minutes per week of moderately intense physical activity.Participants will choose one of the following interventions:
  GLB-GROUP: Individuals who choose group delivery will attend weekly in-person group meetings for 12 weeks, then transition to bi-weekly and monthly meetings. GLB-DVD: Consists of a series of taped sessions of a staged GLB group following a script which was developed to closely follow the original Group Lifestyle Balance. Participants in GLB-DVD will also be invited to attend monthly group meetings and will receive weekly telephone calls from a trained coach.
Period: Overall Study
Arm/Group | Current Intervention | Delayed Intervention
Started | 148 | 75
Completed | 137 | 71
Not Completed | 11 | 4
Not completed — Lost to Follow-up | 7 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Relocated from area | 1 | 2
Not completed — Discontinued Intervention | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Current Intervention: At enrollment, participants are randomly assigned to "Current Intervention" will receive the intervention immediately.The intervention is based on the Diabetes Prevention Program's successful lifestyle intervention with goals of achieving a 7% weight loss, and progressively increasing physical activity to 150 minutes per week of moderately intense physical activity.Participants will choose one of the following interventions:
  GLB-GROUP: Individuals who choose group delivery will attend weekly in-person group meetings for 12 weeks, then transition to bi-weekly and monthly meetings. GLB-DVD: Consists of a series of taped sessions of a staged GLB group following a script which was developed to closely follow the original Group Lifestyle Balance. Participants in GLB-DVD will also be invited to attend monthly group meetings and will receive weekly telephone calls from a trained coach.
- Delayed Intervention: At enrollment, participants are randomly assigned to "Delayed intervention" will receive the intervention in 6 months. The intervention is identical to that received by participants assigned to the Current Intervention Arm and is based on the Diabetes Prevention Program's successful lifestyle intervention with goals of achieving a 7% weight loss, and progressively increasing physical activity to 150 minutes per week of moderately intense physical activity.Participants will choose one of the following interventions:
  GLB-GROUP: Individuals who choose group delivery will attend weekly in-person group meetings for 12 weeks, then transition to bi-weekly and monthly meetings. GLB-DVD: Consists of a series of taped sessions of a staged GLB group following a script which was developed to closely follow the original Group Lifestyle Balance. Participants in GLB-DVD will also be invited to attend monthly group meetings and will receive weekly telephone calls from a trained coach.
- Total: Total of all reporting groups
Arm/Group | Current Intervention | Delayed Intervention | Total
Number analyzed (Participants) | 148 | 75 | 223
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.0 (11.4) | 57.2 (11.6) | 58.4 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 47 | 139
  Male | 56 | 28 | 84
Region of Enrollment [Number; unit: participants]
  United States | 148 | 75 | 223

OUTCOME MEASURES:

1. Primary Outcome: Changes in Weight Between Baseline and Post-intervention (Assessed at 6 Months After Commencement of Intervention) Compared to Delayed Intervention Participants.
Description: Weight was measured twice using a digital physician's scale (DETECTO® PD100) placed on a hard, flat surface. Participants were asked to remove their shoes and stand in the middle of the scale with eyes straight forward and without touching any surface. The participant was asked to step down from the scale between measures. If the measures were more than 0.5 pounds apart, a third measure was taken. Weight is reported in pounds.
Time Frame: Baseline and post-intervention (assessed at 6 months after commencement of intervention)
Population: Intent to treat using last observation carried forward when data are missing.
Measure: Mean (Standard Deviation); unit: Pounds
Arm/Group | Current Intervention | Delayed Intervention
Number analyzed (Participants) | 148 | 75
Pounds | -10.4 (10.1) | -1.8 (7.8)

2. Secondary Outcome: Changes in Fasting Glucose Between Baseline and Post-intervention (Assessed at 6 Months After Commencement of Intervention) Compared to Delayed Intervention Participants.
Description: After the participant signed the consent, they were taken to the private phlebotomy area. The participant sat in a stationary chair and placed their arm of choice for the blood draw flat on the table, on top of the BloodBloc pad. The participant was asked the last time they had anything to eat or drink, including candy, mint, gum, cough drops, cough syrup, coffee or tea, (participants were expected to fast for 8-12 hours prior to their assessment visit). If the participant had anything to eat or drink, other than water, the blood draw was rescheduled. The fasting blood sample was analyzed by Quest Diagnostics™ laboratory for the worksite and community/senior centers.
Time Frame: Baseline and post-intervention (assessed at 6 months after commencement of intervention)
Population: Intent to treat using last observation carried forward when data are missing. Individuals with medication changes related to the outcome were excluded from analysis.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Current Intervention | Delayed Intervention
Number analyzed (Participants) | 148 | 72
mg/dl | -1.9 (8.0) | -1.5 (7.1)

3. Secondary Outcome: Changes in Fasting Insulin Between Baseline and Post-intervention (Assessed at 6 Months After Commencement of Intervention) Compared to Delayed Intervention Participants.
Description: Venous blood draw: After the participant signed the consent, they were taken to the private phlebotomy area. The participant sat in a stationary chair and placed their arm of choice for the blood draw flat on the table, on top of the BloodBloc pad. The participant was asked the last time they had anything to eat or drink, including candy, mint, gum, cough drops, cough syrup, coffee or tea, (participants were expected to fast for 8-12 hours prior to their assessment visit). If the participant had anything to eat or drink, other than water, the blood draw was rescheduled. The fasting blood sample was analyzed by Quest Diagnostics™ laboratory for the worksite and community/senior centers.
Time Frame: Baseline and post-intervention (assessed at 6 months after commencement of intervention)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Current Intervention | Delayed Intervention
Number analyzed (Participants) | 147 | 71
mg/dl | -0.18 (5.1) | 0.81 (5.2)

4. Secondary Outcome: Changes in Fasting Lipids (Total Cholesterol) Between Baseline and Post-intervention (Assessed at 6 Months After Commencement of Intervention) Compared to Delayed Intervention Participants.
Description: Venous blood draw: After the participant signed the consent, they were taken to the private phlebotomy area. The participant sat in a stationary chair and placed their arm of choice for the blood draw flat on the table, on top of the BloodBloc pad. The participant was asked the last time they had anything to eat or drink, including candy, mint, gum, cough drops, cough syrup, coffee or tea, (participants were expected to fast for 8-12 hours prior to their assessment visit). If the participant had anything to eat or drink, other than water, the blood draw was rescheduled. The fasting blood sample was analyzed by Quest Diagnostics™ laboratory for the work site and community/senior centers.
Time Frame: Baseline and post-intervention (assessed at 6 months after commencement of intervention)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Current Intervention | Delayed Intervention
Number analyzed (Participants) | 133 | 67
mg/dl | -2.5 (22.4) | -0.5 (20.9)

5. Secondary Outcome: Changes in Fasting Lipids (Triglycerides) Between Baseline and Post-intervention (Assessed at 6 Months After Commencement of Intervention) Compared to Delayed Intervention Participants.
Description: as for outcome 3
Time Frame: Baseline and post-intervention (assessed at 6 months after commencement of intervention)
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | Current Intervention | Delayed Intervention
Number analyzed (Participants) | 133 | 66
mg/dl | -1.0 [-28 to 19] | 6.5 [-25 to 33]

6. Secondary Outcome: Changes in Fasting Lipids (HDL Cholesterol) Between Baseline and Post-intervention (Assessed at 6 Months After Commencement of Intervention) Compared to Delayed Intervention Participants.
Description: as for outcome 3
Time Frame: Baseline and post-intervention (assessed at 6 months after commencement of intervention)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Current Intervention | Delayed Intervention
Number analyzed (Participants) | 133 | 67
mg/dl | 0.3 (7.6) | -0.6 (6.4)

7. Secondary Outcome: Changes in Fasting Lipids (LDL Cholesterol) Between Baseline and Post-intervention (Assessed at 6 Months After Commencement of Intervention) Compared to Delayed Intervention Participants.
Description: as for outcome 3
Time Frame: Baseline and post-intervention (assessed at 6 months after commencement of intervention)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Current Intervention | Delayed Intervention
Number analyzed (Participants) | 130 | 64
mg/dl | -1.3 (19.1) | -1.8 (20.0)

8. Secondary Outcome: Changes in A1c Between Baseline and Post-intervention (Assessed at 6 Months After Commencement of Intervention) Compared to Delayed Intervention Participants.
Description: Venous blood draw: After the participant signed the consent, they were taken to the private phlebotomy area. The participant sat in a stationary chair and placed their arm of choice for the blood draw flat on the table, on top of the BloodBloc pad. The participant was asked the last time they had anything to eat or drink, including candy, mint, gum, cough drops, cough syrup, coffee or tea, (participants were expected to fast for 8-12 hours prior to their assessment visit). If the participant had anything to eat or drink, other than water, the blood draw was rescheduled. The fasting blood sample was analyzed by Quest Diagnostics™ laboratory for the worksite and community/senior centers. A1c is a measure of glucose control over approximately an 8 to 12 week period.
Time Frame: Baseline and post-intervention (assessed at 6 months after commencement of intervention)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Current Intervention | Delayed Intervention
Number analyzed (Participants) | 148 | 72
percentage of glycosylated hemoglobin | -0.11 (0.16) | -0.01 (0.16)

9. Secondary Outcome: Changes in Systolic Blood Pressure (BP) Between Baseline and Post-intervention (Assessed at 6 Months After Commencement of Intervention) Compared to Delayed Intervention Participants.
Description: Blood pressure was measured in the right arm with the participant seated comfortably with the right arm resting on a table. All participants were asked to rest quietly with feet flat on the floor for five minutes. Following the five minute wait, the radial pulse was measured in the right arm and pulse obliteration level was assessed. The cuff was inflated to the peak inflation rate and the pressure released at a rate of 2mm/Hg per second. First appearance and last heard (phase V) Korotkoff's sounds were utilized to determine systolic and diastolic blood pressure respectively. The cuffed arm was then raised for 5 seconds after each inflation with a wait period of 30 seconds between each blood pressure reading. Blood pressure was repeated twice with the average computed. If it was not possible to measure blood pressure in the right arm, the left arm was utilized and noted in the participant record.
Time Frame: Baseline and post-intervention (assessed at 6 months after commencement of intervention)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Current Intervention | Delayed Intervention
Number analyzed (Participants) | 138 | 71
mmHg | -2.5 (11.2) | 0.6 (9.0)

10. Secondary Outcome: Changes in Waist Circumference Between Baseline and Post-intervention (Assessed at 6 Months After Commencement of Intervention) Compared to Delayed Intervention Participants.
Description: The participant was asked stand with feet together. The waist was measured using a cloth measuring tape around the abdomen. The midpoints were marked horizontally at midpoint between highest point of the iliac crest and lowest part of the costal margin in the mid-axillary line. Both sides of the waist were marked using a cosmetic pencil. The participant was asked to have arms at side and to breathe in, out and hold, and then the measurement was taken. Waist measurement was recorded to the nearest quarter inch. The measure was repeated twice. If waist measures differ by more than one-half inch, a third measurement was recorded.
Time Frame: Baseline and post-intervention (assessed at 6 months after commencement of intervention)
Population: Intent to treat using last observation carried forward when data are missing.
Measure: Mean (Standard Deviation); unit: inches
Arm/Group | Current Intervention | Delayed Intervention
Number analyzed (Participants) | 148 | 75
inches | -1.5 (2.0) | -0.05 (1.8)

11. Secondary Outcome: Changes in Self-reported Physical Activity Between Baseline and Post-intervention (Assessed at 6 Months After Commencement of Intervention) Compared to Delayed Intervention Participants.
Description: The Modifiable Activity Questionnaire (MAQ) was designed by Dr. Kriska. It has been used to assess activity in a variety of populations and age groups over various time frames and was used to assess physical activity levels in the DPP. The MAQ includes both a leisure and an occupational activity section since the homogeneity of energy expenditure related to both of these components of activity within many study populations cannot be assumed. In addition, the MAQ was designed to be modified, based upon pilot testing, prior to its usage, in order to maximize the feasibility and appropriateness of the physical activity instrument to the population of interest. The MAQ has been shown to be both reliable and valid (through comparisons with activity monitors, fitness (field) testing, and the doubly labeled water technique) in adults and adolescents alike. The MAQ has been used to assess a variety of time frames from past year and past week to a lifetime of activity.
Time Frame: Baseline and post-intervention (assessed at 6 months after commencement of intervention)
Population: Intent to treat using last observation carried forward when data are missing.
Measure: Median (Inter-Quartile Range); unit: MET-hrs leisure activity
Arm/Group | Current Intervention | Delayed Intervention
Number analyzed (Participants) | 148 | 75
MET-hrs leisure activity | 13 [2.6 to 28.2] | 6.6 [-0.7 to 17.4]

12. Secondary Outcome: Changes in Diastolic Blood Pressure (BP) Between Baseline and Post-intervention (Assessed at 6 Months After Commencement of Intervention) Compared to Delayed Intervention Participants.
Description: as for outcome 9
Time Frame: Baseline and post-intervention (assessed at 6 months after commencement of intervention)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Current Intervention | Delayed Intervention
Number analyzed (Participants) | 138 | 71
mmHg | -1.3 (8.8) | -1.0 (7.9)

ADVERSE EVENTS:
Time Frame: 1 year for Immediate arm, 1.5 years for Delayed arm.
Groups:
- Current Intervention: No unexpected or unanticipated adverse events occurred in the Current Intervention group.
- Delayed Intervention: No unexpected or unanticipated adverse events occurred in the Delayed Intervention group.
Arm/Group | Current Intervention | Delayed Intervention
Serious Adverse Events (participants affected / at risk) | 0/148 | 0/75
Other Adverse Events (participants affected / at risk) | 0/148 | 0/75

LIMITATIONS AND CAVEATS:
Physical activity data was self-reported. Sample was predominantly white, female, which may not be representative of other groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No